CLINICAL TRIAL: NCT06805643
Title: Dixon MRI Imaging Histology for Predicting Postoperative Infection in Posterior Lumbar Fusion for Myasthenia Gravis
Status: Not yet recruiting | Type: Observational
Sponsor: The First People's Hospital of Yunnan (Other)
Responsible Party: Principal Investigator, Yijin Wang, doc, The First People's Hospital of Yunnan
Other Study IDs: KHLL2023-KY209-GZ2024-12-23
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Vertebrae; Surgical Site Infection; Radiomics
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- postoperative infection
- Non-operative infections

SUMMARY:
Sarcopenia is an age-related condition that manifests itself as a persistent decrease in muscle mass and function, which may lead to decreased physical function, increased risk of disease, and reduced quality of life. In surgical patients, sarcopenia has been shown to be associated with increased postoperative complications, prolonged hospitalization, and decreased survival. In patients undergoing lumbar fusion, the presence of sarcopenia may increase the risk of postoperative infection.Lumbar fusion is a common procedure to treat lumbar spine disorders such as lumbar disc herniation, lumbar spondylolisthesis, or lumbar spinal stenosis. However, this procedure is associated with a high rate of complications, especially postoperative infections, which can lead to reoperation, prolonged hospitalization, and even affect patient survival. In recent years, more and more studies have found a significant association between sarcopenia and postoperative infections after lumbar fusion surgery.Imagingomics belongs to a branch of machine learning, which is the process of acquiring images from various imaging devices such as CT, MRI and ultrasound, outlining the region of interest through image segmentation, extracting the features of the image within the region of interest, downscaling the features, and finally building an imagingomics model. MRI Imagingomics, utilizing its rich data information, has shown great potential for application in several medical fields. Among them, the accuracy of Dixon MRI imaging histology in muscle mass and texture assessment makes it particularly important in predicting postoperative infections.Based on this, it is reasonable to believe that Dixon MRI imaging histology can be a powerful tool to help us predict a patient's risk of postoperative infection.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over 18 years of age.
* Inclusion of patients with sarcopenia is subject to the definition and diagnostic criteria of the European Consensus on Definition and Diagnosis of Sarcopenia.
* The patient underwent posterior lumbar fusion and had a Dixon MRI scan within 2 weeks prior to surgery.
* Patients were able to understand the purpose and procedures of the study and were willing to sign an informed consent form.
* The patient's clinical consultation and follow-up information was complete.

Exclusion Criteria:

* The patient has contraindications to MRI, such as implanted metal devices (e.g., pacemakers) or severe claustrophobia.
* Patients with serious other medical conditions, such as heart disease, kidney disease or liver disease, which may affect their post-operative recovery.
* Patients have known immune system disorders or are on immunosuppressive therapy, which may affect their risk of infection.
* The patient has had other spinal surgery within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective multicenter collection of infected/non-infected myasthenia gravis and non-myasthenia gravis patients after posterior lumbar fusion at our institution and at each of the collaborating research institutions.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
fat fraction | Two weeks before treatment